CLINICAL TRIAL: NCT02560376
Title: 68Ga-NOTA-exendin-4 PET/CT for the Localization of Insulinoma and Diagnosis of Nesidioblastosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM12; ZIAEB000073 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-05

CONDITIONS: Insulinoma; Nesidioblastosis
Keywords: PET/CT; glucagon-like peptide-1 receptor (GLP-1R) imaging
MeSH Terms: conditions — Insulinoma; Nesidioblastosis | interventions — 68Ga-NOTA-exendin-4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-exendin-4 PET/CT (Experimental): The patients were injected with 55.5-111 MBq of 68Ga-NOTA-exendin-4 PET/CT in one dose intravenously and underwent PET/CT scan 30-60 min later.
  Interventions: Drug: 68Ga-NOTA-exendin-4

INTERVENTIONS:
Drug: 68Ga-NOTA-exendin-4 — 68Ga-NOTA-exendin-4 were injected into the patients before the PET/CT scans
  Other Names: 68Ga-NOTA-MAL-cys40-exendin-4

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-exendin-4 in insulinoma and nesidioblastosis patients. A single dose of 55.5-111 Mega-Becquerel (MBq) 68Ga-NOTA-exendin-4 will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
68Ga-NOTA-exendin-4 is an optimal probe targeting GLP-1R. The investigators will determine the use of 68Ga-NOTA-exendin-4 PET/CT in the detection of insulinomas, and to compare its diagnostic value with conventional imaging. GLP-1R imaging, specifically expressed on pancreatic beta cell surface, might help with diagnosis of different types of nesidioblastosis (ie. focal or diffuse type), and may improve the treatment strategy of nesidioblastosis. The investigator will determine the use of 68Ga-NOTA-exendin-4 PET/CT in differentiating nesidioblastosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypoglycaemia in the presence of neuroglycopenic symptoms and documented Whipple's triad.
* Biochemically proven endogenous hyperinsulinemic hypoglycaemia (plasma glucose concentration <3.0 mM, insulin >3 µU/ml, and C-peptide >0.6 ng/ml).
* Conventional imaging within 1 month
* Signed written consent
* Age above 6 years (congenital hyperinsulinemic with the symptoms onset in school age is also the subject of this study)

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Renal function: serum creatinine > 3.0 mg/dl
* Known allergy against exendin-4
* Any medical condition that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-exendin-4 PET/CT in Diagnosis of Insulinoma and Nesidioblastosis | 1 year

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China